CLINICAL TRIAL: NCT01503099
Title: Intestinal Tuberculosis Diagnostics and the Differentiation From Crohn's Disease in Populations of High vs. Low Tuberculosis Endemicity
Brief Title: Intestinal Tuberculosis Diagnostics and the Differentiation From Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government); The Unger-Vetlesen Medical Fund, Jersey, C.I (Unknown); Odd Fellow Medical Fund, Norway (Unknown)
Responsible Party: Bjorn Moum, Oslo University Hospital, Aker
Other Study IDs: LDS 150
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Intestinal Tuberculosis; Pulmonary Tuberculosis; Crohn's Disease
Keywords: ITB; PTB; CD
MeSH Terms: conditions — Tuberculosis, Pulmonary; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples frozen at -20'C. Blood serum samples frozen at -20'C. Saliva samples stored at room temperature. Paraffin embedded intestinal biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Active ITB: Patients with active intestinal tuberculosis (ITB)
- Controls India: Healthy subjects serving as controls
- CD India: Patients with active Crohn's Disease (CD) in India
- Active PTB: Patients with active pulmonary tuberculosis (PTB)
- CD Norway: Patients with active Crohn's Disease (CD) in Norway
- Controls Norway: Healthy subjects serving as controls in Norway

SUMMARY:
One aims to devise a method for the screening and differentiation of intestinal tuberculosis and Crohn's Disease. Additionally, one aims to detect and survey multidrug resistant TB.

DETAILED DESCRIPTION:
Intestinal tuberculosis (ITB) and Crohn's disease (CD) may present identically; the consequence of misdiagnosing and mistreating one disease for the other may be grave. CD is on the increase worldwide while TB re-emerges in areas of low TB endemicity. Current diagnostic guidelines evolve from research in areas with low TB prevalence, thereby being inappropriate in TB endemic regions. To date, no simple or non-invasive methods exist to diagnose ITB and to differentiate it from CD.

One aims to devise a method for screening and differentiation of the two diseases. By using non-invasive rapid tests one wishes to make diagnostics available to resource poor settings. Ideally, referrals to invasive diagnostic procedures would decrease, thus liberating economic and staff resources. Furthermore, patients may avoid unnecessary, expensive and often inconclusive advanced procedures. Additionally, one aims to detect and survey multidrug resistance caused by empiric TB treatment, which in itself obscures ITB diagnosis.

This case control study matches 50 ITB patients and 50 CD patients with 100 healthy controls in India, and 50 CD patients with 100 healthy controls in Norway. Comparative statistical analysis will be carried out. Challenges include patient adherence and sample handling. Non-TB gastrointestinal infections may confound the results and will be adjusted for.

Recently published data suggests that the serum/faecal calprotectin ratio may be used to discriminate ITB from healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age.
* ITB as per standard criteria a), and one or more of b) to e) must be fulfilled (Gold standard):

  1. Endoscopic apparent intestinal tuberculosis: transverse ulcers, pseudopolyps, involvement of fewer than four intestinal segments, patulous ileo-coecal valve
  2. Histological evidence of tubercles/granulomas with caseation necrosis in intestinal biopsies
  3. DNA of M.tb detected by PCR of intestinal biopsies
  4. Positive immunohistochemistry in intestinal biopsies.
  5. Histological demonstration of acid fast bacilli in a lesion.
* Active Crohn's disease as per standard criteria (Gold standard), at least two of the following:

  1. Clinical: inflammatory, perforating (fistulising) disease, obstructive symptoms secondary to small bowel stenosis or stricture.
  2. Endoscopic: deep linear or serpingenous ulcerations, discrete ulcers in normal appearing mucosa, cobble-stoning or discontinuous or asymmetrical inflammation.
  3. Radiographic: segmental disease (skip lesions), small bowel or colonic strictures, stenosis or fistula.
  4. Histological: sub-mucosal or transmural inflammation, granulomas, focal cryptitis and chronic inflammatory infiltration, skip lesions including rectal sparing (no topical rectal therapy).

Exclusion Criteria:

a) Age below 18 years b) HIV positive c) Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients from four secondary or tertiary care referral centres in the two southernmost states in India (Kerala and Tamil Nadu).
  Consecutive patients from nine secondary or tertiary care referral centres in South-East Norway.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Calprotectin levels in patients with active intestinal tuberculosis | 18 months
  Establishment of serum and faecal calprotectin levels in patients with active intestinal tuberculosis in comparison with healthy control subjects, patients with Crohn's Disease and patients with active pulmonary tuberculosis.

SECONDARY OUTCOMES:
Levels of calprotectin in patients with intestinal tuberculosis after antituberculous therapy. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Moum, M.D Ph.D, Study Chair — Oslo University Hospital, Aker; Gunnar Bjune, M.D Ph.D, Study Chair — University of Oslo, Dept. of International Health
Locations (2):
- Population Health & Research Institiute, Medical College, Trivandrum, Kerala, India
- Lovisenberg Diakonal Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Larsson, G; Shenoy, KT; Roseth, A; Bjune, G; Moum, B. Diagnosis and differentiation of intestinal tuberculosis and Crohn's disease by use of faecal and serum calprotectin. INFLAMMATORY BOWEL DISEASES 17: S35-S35 Suppl. 1 JAN 2011